CLINICAL TRIAL: NCT05687227
Title: The Effect on Women's Attitude and Anxiety Levels Regarding Gynecological Examination of Online Education and Counseling
Brief Title: Online Education and Counseling Regarding Gynecological Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Belma Toptas Acar, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BELMA TOPTAŞ ACAR
Record Dates: First submitted 2022-10-02; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Gynecological Disease
Keywords: gynecological examination; attitude; anxiety; online; education; counseling
MeSH Terms: conditions — Genital Diseases, Female; Behavior; Anxiety Disorders | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENT GROUP (Experimental): The trainings were held in groups of 4-6 people. The trainings, which were held in three sessions, were held on the days and times that were convenient for the participants. Since the participants were required to attend all sessions, additional session/sessions were held in case of not being able to attend the trainings. Participants in the control and experimental groups were called and the day they would come for the control was determined, and they went to the gynecology outpatient clinic. The post-test questionnaire was applied to the participants in the control and experimental groups in the first 3 months. Until the end of the research, the participants were told that they could reach the researcher at any time and ask questions. Finally, at the 6th month, a post-test form was applied to the participants.
  Interventions: Behavioral: Online education and counseling
- CONTROL GROUP (No Intervention): No training or counseling was given to the control group. Participants in the control and experimental groups were called and the day they would come for the control was determined, and they went to the gynecology outpatient clinic. The post-test questionnaire was applied to the participants in the control and experimental groups in the first 3 months. Finally, at the 6th month, a post-test form was applied to the participants.

INTERVENTIONS:
Behavioral: Online education and counseling — Online education and counseling regarding gynecological examination
  Arms: EXPERIMENT GROUP

SUMMARY:
This research was carried out to determine the effect of online education and counseling on women's attitudes and anxiety levels regarding gynecological examination.

The research is a pre-test-post-test, randomized controlled experimental study.

DETAILED DESCRIPTION:
The research is a pre-test-post-test, randomized controlled experimental study. Simple randomization method was used to assign the participants to the groups. The sample consisted of a total of 100 women (experimental group: 50 women and control group: 50 women). The study was carried out with women who applied to Aydın Adnan Menderes University Application and Research Hospital, Gynecology Clinic, Gynecology Outpatient Clinic and met the study criteria.

ELIGIBILITY:
Inclusion Criteria:

* Applying to Aydın Adnan Menderes University Application and Research Hospital, Gynecology Clinic, Gynecology Clinic,
* Coming to the examination within the first 3 months after the examination,
* Internet access,
* Having a Whatsapp or e-mail address,
* Able to read and write,
* Able to speak and understand Turkish,
* Women in the 18-50 age group are included.

Exclusion Criteria:

* Having a communication (speech, hearing, etc.) disability,
* Having any psychological illness,
* Pregnant and postpartum,
* Diagnosed with cancer,
* Women who received infertility diagnosis and treatment were excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
A pre-test was applied to 100 women constituting the sample of the study. | up to 9 months.
  Before the online training and counseling, a pre-test was applied to a total of 100 participants, 50 of which were in the experimental group and 50 in the control group. In the pre-test question form created by the researcher in the light of the literature, sociodemographic (questions 1-9), obstetrics (questions 10-13), gynecological characteristics (questions 14-23) and attitudes towards gynecological examination (16 questions ).
The State and Trait Anxiety Inventory was applied to 100 women constituting the sample of the study. | up to 9 months.
  The State and Trait Anxiety Inventory, which was developed by Spielberger (1970) and adapted to Turkish by Öner and Le Compte in 1983, was used. The first 20 questions in the scale measure "state anxiety" and the next 20 questions measure "trait anxiety". A score of 0-19 indicates no anxiety. While 20-39 indicates mild anxiety, 40-59 moderate and 60-79 severe anxiety, 80 points are considered as panic. The minimum value to be taken from the state anxiety scale is "0" and the maximum value is "80". The minimum value to be taken from the trait anxiety scale is "0" and the maximum value is "80". As the score increases, the level of anxiety also increases.

SECONDARY OUTCOMES:
The posttest was applied to 68 people who were pretested within the first 3 months after the pretest was applied. | The pre-test implementation phase was completed in 9 months. This process took a total of 1 year, since the last test was applied to the last participants within the 3rd month.
  Online training and counseling about gynecological examination was applied to the experimental group. No counseling or training was given to the control group. Trainings on gynecological examination were carried out in 3 sessions by determining the days and hours that women are suitable for via Google Meet. The trainings were carried out in groups of 4-6 people. The women in the experimental and control groups who will come for the examination were reached in advance and information was obtained about when they would come, and they went to the gynecology outpatient clinic on the day they would come for the check-up. The post-test form was applied to the participants face to face and the form was filled by the participant himself. The post-test form included attitude questions about gynecological examination.
The State and Trait Anxiety Inventory was applied to 68 people who were pretested within the first 3 months after the pretest was applied. | The pre-test implementation phase was completed in 9 months. This process took a total of 1 year, since the last test was applied to the last participants within the 3rd month.
  The State and Trait Anxiety Inventory, which was developed by Spielberger (1970) and adapted to Turkish by Öner and Le Compte in 1983, was used. The first 20 questions in the scale measure "state anxiety" and the next 20 questions measure "trait anxiety". A score of 0-19 indicates no anxiety. While 20-39 indicates mild anxiety, 40-59 moderate and 60-79 severe anxiety, 80 points are considered as panic. The minimum value to be taken from the state anxiety scale is "0" and the maximum value is "80". The minimum value to be taken from the trait anxiety scale is "0" and the maximum value is "80". As the score increases, the level of anxiety also increases.

OTHER OUTCOMES:
Filling in the second post-test questionnaire online in the 6th month after both groups filled out the pre-test questionnaire. | Since the second posttest form was 3 months after the first posttest form (6 months after the pretest questionnaire), this process was completed in the 15th month from the beginning of the study in total.
  Online training and counseling about gynecological examination was applied to the experimental group. No counseling or training was given to the control group. The post-test form was applied to the participants online. The same questions regarding the gynecological examination included in the posttest questionnaire, which must be completed within the first 6 months after the pretest is completed.
The State and Trait Anxiety Inventory was administered again in the 6th month to 68 people who were posttested in the first 3 months. | Since the second posttest form was 3 months after the first posttest form (6 months after the pretest questionnaire), this process was completed in the 15th month from the beginning of the study in total.
  The first 20 questions in the scale measure "state anxiety" and the next 20 questions measure "trait anxiety". A score of 0-19 indicates no anxiety. While 20-39 indicates mild anxiety, 40-59 moderate and 60-79 severe anxiety, 80 points are considered as panic. The minimum value to be taken from the state anxiety scale is "0" and the maximum value is "80". The minimum value to be taken from the trait anxiety scale is "0" and the maximum value is "80". As the score increases, the level of anxiety also increases

CONTACTS AND LOCATIONS:
Overall Officials: BELMA TOPTAŞ ACAR, Res.assist, Principal Investigator — belma.toptas@adu.edu.tr
Locations (1):
- Aydın Adnan Menderes University Application and Research Hospital, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I have completed the data of my doctoral thesis. There were 37 experimental groups and 31 controls who completed the study to the end. I wrote my thesis. After making the necessary arrangements with my advisor, I will have my thesis defense exam in December 2022. I will share the summary of my thesis within the month after the defense.
Supporting Information: CSR
Time Frame: January 2023- December 2024
Access Criteria: Klinik Çalışma Raporu (KSS)